CLINICAL TRIAL: NCT03256604
Title: A Sputum Screening Test to Rule-out Pneumonia at an Early Stage
Acronym: self-test
Status: Completed | Type: Observational
Sponsor: University Hospital, Linkoeping (Other)
Collaborators: Linkoeping University (Other Government); PEAS Institut (Unknown)
Responsible Party: Principal Investigator, Fariba Nayeri, PhD, MD, associated professor, University Hospital, Linkoeping
Other Study IDs: Dexact-resp
Record Dates: First submitted 2017-08-16; First posted 2017-08-22 (Actual); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Pneumonia; Community-acquired Pneumonia; Exacerbation Copd
Keywords: point of care, HGF, innate immunity
MeSH Terms: conditions — Pneumonia; Community-Acquired Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Sputum samples from all included cases are kept frozen -70 C coded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Fresh left-over sputum: All fresh sputum samples that were sent to the Department of Microbiology between November 1 2015 and January 30 2016 under the standard requirements for sputum cultures at the accredited (ISO 17025 and 15189 beginning in 1993) laboratory were kept cold (4-8 ͦC) after analysis by microscope and cultures until it was collected and coded by the study nurse in the evening (left-over samples).
  Interventions: Diagnostic Test: left-over sputum

INTERVENTIONS:
Diagnostic Test: left-over sputum — Totally 467 samples were gathered from different clinics, and the diagnostic procedures and the therapeutic approaches were completely unknown to the study group. The coded samples were stored at 4-8°C and analyzed within 72 hours of sampling using the sputum strip test. From April to June 2016, a physician and the study nurse reviewed the journals. The age, sex, length of stay on ward, the clinical symptoms, the blood and sputum cultures and PCR along with the results, the X-rays, the antibiotic therapy, CRB-65 and the ultimate diagnosis code (ICD-10) were documented in Excel-files.

SUMMARY:
In patients with clinical symptoms of respiratory infection, rapid identification of cases requiring antibiotic therapy is crucial to avoid development of multiple resistant bacteria. Identification of local acute-phase reactants can help assess the host's response to bacterial infection at the injury site. Here, the investigators developed an affordable, stable, feasible, and accurate diagnostic tool based on a locally produced protein with specific binding affinity to polysaccharides. The investigators further evaluated the ability of the novel test strip to rule out pneumonia.

DETAILED DESCRIPTION:
A lower respiratory tract infection is a serious situation that can abruptly become complicated by sepsis, respiratory failure, lung tissue necrosis, and multiple organ dysfunction. Hence, empiric antibiotic treatment is commonly initiated as soon as infection is suspected and cultures and/or other diagnostic tests are procured, representing a major reason for antibiotic prescription. Widespread antibiotic overuse and misuse have led to the emergence of multiple resistant bacterial strains, posing a major health threat. There exists a critical need for practical solutions to prevent antibiotic overuse, especially in communities where antibiotics are available without prescription.

Pathophysiologic studies show that infection does not result from bacterial or viral overgrowth alone, but rather from the microorganisms' penetration beyond the host immune system. Therefore, infection assessment requires investigation of both microorganism presence and the defense mechanisms activated within the patient's body. Bacteria overgrowth leads to lung tissue inflammation, recruitment of white blood cells to the infected area, and chemokine and cytokine production and release, which can cause the alveoli to become filled with fluid, leading the patient to develop a cough with phlegm or pus, fever, chills, and dyspnea.

Microbiological diagnosis of lower respiratory tract infections requires assessment of the invading microorganism by examination of sputum using microscopy, quantitative culture, and PCR. However, such microbiological investigations have limited value in pneumonia management. Polymicrobial flora make it difficult to interpret cultures from patients with chronic bronchitis. It is also difficult to evaluate cultures from nosocomial pneumonia since the pathogenic bacteria are often identical to those appearing in the throat flora. Immunosuppressed patients frequently produce sputum containing low number of white blood cells. The patient's clinical signs, such as respiratory and circulatory status, are the most reliable markers for determining treatment efficacy.

In practice, most physicians choose to examine additional markers at early stages to closely monitor the effects of therapy, particularly in high-risk patients who have been admitted to intensive care units. Commonly used systemic markers include body temperature, C-reactive protein (CRP), procalcitonin (PCT), and interleukin 6 (IL-6). Hepatocyte growth factor (HGF) concentration reportedly increases during organ damage, such as that caused by infectious diseases. Studies show increased HGF concentrations in serum and exhaled-breath condensate from patients with pneumonia, with HGF presence being significantly correlated with survival. Moreover, HGF levels markedly decrease within 48 hours of initiating appropriate antibiotic therapy. Surface plasmon resonance (SPR) results indicate that HGF produced during acute infection shows high affinity for the extracellular matrix component heparan sulfate proteoglycan (HSPG). These findings suggest that HGF assessment in sputum could be a tool for detecting bacterial infection at the site of injury.

Proteins can be detected based on their specific interaction with a corresponding antibody. However, this measurement system relies on specialized resources, limiting its usefulness in non-equipped centers or as a self-test. Metachromasia is a characteristic color change exhibited by certain aniline dyes upon binding to chromotropic substances. This phenomenon has been widely used in histology. Methylene blue (O-Toluidine) is an excellent metachromatic dye that changes from blue to pink upon binding to high-molecular-weight polysaccharides, such as sulfated glycan. The pink dye will then quickly turn back to blue following addition of a proportional amount of a protein with high affinity to sulfated glycan (inverted metachromacia).

Here the investigators used this approach to develop a new strip test-referred to herein as the index text-to assess the presence of dextran-sulfate-binding proteins in sputum. The investigators then assessed the accuracy of this strip test for detecting bacterial infection in sputum, by analyzing leftover sputum samples that were sent for examination to the Department of Microbiology, University hospital in Linköping.

ELIGIBILITY:
Inclusion Criteria:

* Sputum samples collected for routine diagnostic and reached the laboratory within 12 hours after Collection and considered as representative by microscopy and kept 4-8 C after Culture.

Exclusion Criteria:

* Samples not collected as above

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All cases that searched the open Health care specialist facility at Linkoeping University hospital or were admitted to the ward at different clinics at the University Hospital in Linkoeping between 1st November 2015 to 30th January 2016 due to suspected respiratory infection and sputum samples were collected to be cultured at the Department of Microbiology University Hospital in Linkoeping.
Sampling Method: Probability Sample
Enrollment: 467 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2016-02-05 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Negative predictive value to rule-out pneumonia | Within two years
  The sputum samples were collected randomly without knowledge about the patient or the ultimate diagnosis. The diagnoses were established first after the patient was dismissed from the clinic.
  RESPIRATORY INFECTION Pneumonia The following criteria were used to define pneumonia diagnosis
  1. Clinical signs and symptoms
  2. Changes detected by recent chest radiography
  3. Received antibiotic therapy, irrespective previous antibiotic consumption.
  4. The ultimate diagnosis J13-J18-J690 (ICD-10). Community-acquired pneumonia: The patients without previous respiratory disease.
  Hospital acquired (Nosocomial) pneumonia: Patients (n=11) acquired pneumonia at the hospital at least 48-72 hours after being admitted.

SECONDARY OUTCOMES:
Correlation to HGF and S100A8-A9 (Calprotectin) concentration (Elisa) in sputum | The samples were kept frozen after sampling -20 C and then thawed after 4 months and analyse was performed within 1 day.
  We assessed immunoreactive human HGF and calprotectin (Human S100A8/S100A9 heterodimer) concentrations by ELISA (80 randomly chosen samples) using commercially available ELISA kits (Quantikine ELISA; R&D systems, Inc., Minneapolis, MN, USA). This method measures HGF and calprotectin in serum, plasma, culture media, and other biological fluids. Sputum samples that had been stored -20C were thawed and centrifuged at 1000 g for 10 minutes prior to analysis. The minimum detectable dose (MDD) as defined by supplier for this assay was 0.04 ng/ml for HGF and 0.086 ng/ml for calprotectin.
Correlation to binding affinity to the parts of HGF molecule by Surface plasmon resonance | in 47 samples paired Elisa and SPR analysis was performed on samples kept in -20 C within 4 months after sampling..
  Paired analysis was performed on 47 randomly chosen samples. Measurements and ligand immobilization procedures were conducted using a Biacore 2000 system (GE Healthcare Bio-Sciences AB, Uppsala, Sweden). Three different ligands were immobilized in separate channels on the SPR-chip. The ligands were affinity purified polyclonal antibodies directed against HGF peptides mapping at the N-terminus of human HGFβ (N-19), the N-terminus of human HGFα (N-17), and amino acids 32-176 of human HGFα (H-145). These ligands were diluted 1:10 in 10 mM acetate buffer (pH 4.5) and immobilized to carboxymethylated dextran CM5 chips

OTHER OUTCOMES:
The management routine for pneumonia at Infectious clinic in Linkoeping in last decades | The data was obtained from paper journals from patients that were admitted (December to March) to the Department of Infectious diseases in Linköping in 1970,1980 and1990
  We studied the archived paper journals from patients that were admitted to our ward and dismissed under diagnosis pneumonia/bronchopneumonia, beginning in 1970. We aimed to identify the diagnostic approaches that were used at the same center and had an impact on the correct diagnosis of pneumonia. Patients received a code depending on the date of admission to the ward from January-December and were registered under the code in a book. The codes belonging to a particular diagnosis were collected on a card and kept separately in boxes (one card corresponded to one diagnosis and one year). We randomly chose the first 40 coded cases with a diagnosis of Pneumonia (ICD-9 diagnosis code 486.9) in 1970, 1980, and 1990 and collected the paper journals and identified the criteria for diagnosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Infectious Diseases, Linköping, Östergotland, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Information regarding the samples that were included in statistic calculations, excluded cases with infection, pneumonia 1970-1980-1990, the actual cost of tests performed at our centre for diagnosis of pneumonia and the volunteers joining the feasibility test in Tables A-L
Supporting Information: Study Protocol, ICF, CSR
Time Frame: The data is available and awaiting the URL address to be defined.